CLINICAL TRIAL: NCT01730144
Title: Elucidation of the Mucosal Immune Responses to Live Attenuated Influenza Vaccine In Healthy Adults
Brief Title: Studying Cell Immune Responses to a Live Flu Vaccine in Healthy Adults
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130020; 13-I-0020
Record Dates: First submitted 2012-11-17; First posted 2012-11-21 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-07-12

CONDITIONS: Normal Physiology
Keywords: Nasal Spray Vaccine; Nasal Cells

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Background:

- One form of the influenza vaccine is a nasal spray. It uses a live but weakened flu virus. Researchers want to better under how the live vaccine interacts with the body s immune system. They will test the nasal spray flu vaccine (called FluMist) against a saline (salt water) nasal spray. They will then look at blood and nasal cell samples to see how the vaccine affects these cells immune response.

Objectives:

- To look at immune changes in nasal and blood cells in people who receive live flu vaccine.

Eligibility:

- Healthy volunteers between 18 and 49 years of age.

Design:

* Participants will have five outpatient visits for this study. Each visit will last up to 2 hours.
* At the first visit, participants will have a physical exam and medical history. They will give blood and urine samples. Nasal cell samples will also be collected.
* A week later, participants will have either the nasal spray flu vaccine or a saline spray. They will know which spray they will receive. Blood samples will be collected.
* Two days after the vaccination, they will have another physical exam. Blood and nasal cell samples will be collected.
* At the final two visits (1 week and 1 month after the vaccination), more blood samples will be collected.
* Those who had the saline spray will be able to have the actual vaccine spray at the last study visit.
* The ratio of participants who receive vaccine to those who receive saline will be 4:1.

DETAILED DESCRIPTION:
Two types of influenza vaccines are currently licensed in the US, trivalent inactivated vaccine (TIV), administered by intramuscular injection, and LAIV, administered by nasal spray. Both vaccines are safe and effective in their approved age groups. Neutralizing antibody in the serum has been found to be a correlate of protection for TIV, but the immune correlates of protection for LAIV are not known. Defining the origin and nature of transcriptional responses to LAIV in URT in infected and bystander epithelial and lymphocyte cells in healthy adults will be a highly informative first step in a systems approach toward understanding the molecular basis of viral replication restriction and the regulation of the local mucosal immune responses following LAIV administration.

This natural history study will use a systems biology approach to identify LAIV replication niches among a variety of URT cell types and characterize the host immune response to LAIV. Healthy volunteers aged 18-49 years will be prescreened for low (<1:10) serum HAI titer against the component influenza vaccine virus strains (influenza A H1N1 and H3N2, and influenza B) of the licensed seasonal LAIV. Ten HAIlow or -negative individuals will be vaccinated intranasally with LAIV (n=8) or will receive saline intranasally (n=2). One week prior to and 2 days after vaccine administration, an NP specimen will be collected using flocked NP swabs. A blood sample will be collected at the time of NP swabbing and on Days 7 and 28 after vaccination. Total subject participation time from enrollment/baseline to the final study visit will be 5 weeks.

We propose to recover cells from NP swab samples and sort individual cells of different subsets based on specific surface phenotypic markers. We will then utilize microfluidics-based real-time reverse transcriptase polymerase chain reaction (rRT-PCR) to quantify transcripts from bulk and single cells. These transcripts will include strand-specific influenza RNA for determining virus replication, genes for assigning cells to specific epithelial or lymphocyte subpopulations, selected genes in the IFN signaling pathways to determine innate immune responses, and genes involved in activation and effector functions of different immune cell subsets. Results will be analyzed with several bioinformatics tools, with an emphasis on the differential signaling responses between various cells types. The mucosal transcriptional data will be correlated with B and T cell immunity markers and traditional serology (HAI and neutralization assays) before and after vaccination to identify key factors affecting the immune response to LAIV.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult males and females between 18 and 49 years of age.
* Females of child-bearing potential must have a negative serum beta-human choriogonadotropin (HCG) on Day -7 and agree to use an effective birth control method for the duration of the study (for example, pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; intrauterine device; abstinence from heterosexual intercourse, surgical sterilization). All female subjects will be considered being of child-bearing potential except those who have undergone hysterectomy and those in whom menopause occurred at least 1 year prior to the study.
* General good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator.
* Agree to storage of blood, NP swab, and RNA specimens for future research.
* Available for the duration of the study. Subjects must be willing and able to make follow-up visits as specified by the protocol.

EXCLUSION CRITERIA:

* Any contraindiciations for adults for the receipt of LAIV:

  --Hypersensitivity to eggs, egg proteins, gentamicin, gelatin, or arginine,or life-threatening reactions to previous influenza vaccination.
* Currently breast-feeding.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urine testing. Clinically significant alanine aminotransferase (ALT) levels, as determined by one of the protocol investigators will be exclusionary at baseline, prior to vaccination.
* Evidence of upper respiratory tract illness (URI) including fever, sore throat, and rhinorrhea. Enrollment of subjects with evidence of URI on Study Day -7 will be temporarily deferred.
* Deviated nasal septum or nasal obstruction.
* Body Mass Index greater than 35.
* NIH employee involved in direct patient care, consistent with the NIH CC policy that employees should avoid patient care for 5 days following receipt of LAIV. In addition, NIH employees must not be under the supervision of the study principal or associate investigators.
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
* Seropositive to the influenza A component viruses of seasonal LAIV (serum HAI titer of greater than or equal to 1:10).
* Has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the study or would render the subject unable to comply with the protocol.
* History of anaphylaxis.
* Current diagnosis of asthma or reactive airway disease (within the past 2 years).
* History of Guillain-Barr(SqrRoot)(Copyright) Syndrome.
* Positive enzyme-linked immunosorbent assay (ELISA) and confirmatory Western blot tests for human immunodeficiency virus-1 (HIV-1).
* Positive ELISA and confirmatory test (e.g., recombinant immunoblotassay) for hepatitis C virus (HCV).
* Positive hepatitis B virus surface antigen (HBsAg) by ELISA.
* Known immunodeficiency syndrome.
* Use of oral, injected, or inhaled corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to enrollment in the study.
* Use of any herbal supplement 30 days prior to study enrollment.
* Receipt of 2012-2013 influenza vaccine (TIV or LAIV).
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to enrollment in the study.
* History of a surgical splenectomy.
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination.
* Current smoker.
* Travel to the Southern Hemisphere 30 days prior to study enrollment or anticipated travel to the Southern Hemisphere during the study.
* Travel on a cruise ship 30 days prior to study enrollment or anticipated travel on a cruise ship during the study.
* Receipt of another investigational vaccine or drug within 30 days prior to enrollment in the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11-17; Primary Completion 2013-04-17 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Significant differences in transcription of selected genes in nasal mucosal epithelial and immune cells isolated from recipients of LAIV compared to pre-vaccination levels in the same cell populations isolated. | One week prior to and 2 days after vaccine administration and on Days 7 and 28 after vaccination.

SECONDARY OUTCOMES:
1) Development of serum antibody assessed by either HAI or microneutralization (MN) assays.2) Development of 200 influenza-specific interferon-gamma (IFN- >=)-secreting cells per million lymphocytes as assessed by enzymelinked immunospo... | One week prior to and 2 days after vaccine administration, and on Days 7 and 28 after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Tara N Palmore, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sen A, Rothenberg ME, Mukherjee G, Feng N, Kalisky T, Nair N, Johnstone IM, Clarke MF, Greenberg HB. Innate immune response to homologous rotavirus infection in the small intestinal villous epithelium at single-cell resolution. Proc Natl Acad Sci U S A. 2012 Dec 11;109(50):20667-72. doi: 10.1073/pnas.1212188109. Epub 2012 Nov 27. PMID 23188796
- [Background] Nakaya HI, Wrammert J, Lee EK, Racioppi L, Marie-Kunze S, Haining WN, Means AR, Kasturi SP, Khan N, Li GM, McCausland M, Kanchan V, Kokko KE, Li S, Elbein R, Mehta AK, Aderem A, Subbarao K, Ahmed R, Pulendran B. Systems biology of vaccination for seasonal influenza in humans. Nat Immunol. 2011 Jul 10;12(8):786-95. doi: 10.1038/ni.2067. PMID 21743478
- [Background] Zhu W, Higgs BW, Morehouse C, Streicher K, Ambrose CS, Woo J, Kemble GW, Jallal B, Yao Y. A whole genome transcriptional analysis of the early immune response induced by live attenuated and inactivated influenza vaccines in young children. Vaccine. 2010 Apr 1;28(16):2865-76. doi: 10.1016/j.vaccine.2010.01.060. Epub 2010 Feb 12. PMID 20153794